CLINICAL TRIAL: NCT06449118
Title: The Effect of Mindfulness Based-stress Reduction Program Applied to Parents With Physically Disabled Children on Stress and Quality of Life: A Single-Blind Randomized Controlled Trial
Brief Title: Effectiveness of Mindfulness-based Stress Reduction Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: c.taskaya
Record Dates: First submitted 2024-05-27; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Stress
Keywords: Mindfulness Stress Reduction Program; physically disabled; parent; quality of life; stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Stress Reduction (Active Comparator): Mindfulness Stress Reduction Program
  Interventions: Behavioral: Mindfulness Stress Reduction Program
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Mindfulness Stress Reduction Program — Mindfulness based-Stress Reduction Program an 8-week program
  Arms: Mindfulness Stress Reduction

SUMMARY:
Having a physically disabled child presents serious challenges for parents, not only in the practice of daily living, but also on a psychological and emotional level. In addition to meeting the constant and complex needs of their children, these parents must also maintain their own emotional balance and psychological well-being. In the long term, high stress levels can seriously compromise parents' mental health and reduce their overall quality of life. Therefore, the development of effective stress management strategies and psychological support mechanisms for parents is critical not only for individual well-being but also for the health of family relationships. Mindfulness practices, in this context, emerge as powerful tools with the potential to increase parents' ability to cope with stress and improve emotional well-being. Therefore, this study aims to determine the effect of the mindfulness stress reduction program applied to parents of physically disabled children on stress and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being able to read and write
* Having a child diagnosed with a physical disability

Exclusion Criteria:

* Having more than one physically disabled child

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Mindful Attention Awareness Scale | Two months
  Mindful Attention Awareness Scale(MAAS), measures the general level of awareness of and attentiveness to current processes in daily life. The scale is a six-point Likert-type scale consisting of 15 items. The scale is a 6-point Likert scale including almost always (1), most of the time (2), sometimes (3), rarely (4), very rarely (5), and almost never (6). The MAAS is single-factor and a single total score is obtained from the scale. The lowest score that can be obtained from the scale is 15 and the highest is 90. The higher the score obtained from the scale, the higher the mindfulness level of the individual.
Parent Stress Scale | Two months
  It is a scale developed to measure the stress experienced by parents in their relationships with their children in daily life. The scale is a one-dimensional scale consisting of 16 items. It is a four-point Likert-type scale with the options "always, often, sometimes and never".
World Health Organization's Quality of Life (WHOQOL-BREF) Questionnaire | Two months
  The scale consists of 27 questions in total. This scale, which is completed by the participants, evaluates quality of life from 4 dimensions: physical health domain, psychological domain, social relations domain and environmental domain.